CLINICAL TRIAL: NCT00665665
Title: Safety, Efficacy, Tolerability and Pharmacokinetics of NNC 0070-0002-0182 in Overweight or Obese Healthy Male and Female Volunteers
Brief Title: Safety, Efficacy, Tolerability and Pharmacokinetics of NNC 0070-0002-0182 in Overweight or Obese Male and Female Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial is terminated due to re-evaluation of the compound
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9112-1846
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental)
  Interventions: Drug: NNC 0070-0002-0182; Drug: placebo
- B (Experimental)
  Interventions: Drug: placebo; Drug: NNC 0070-0002-0182
- C (Experimental)
  Interventions: Drug: placebo; Drug: NNC 0070-0002-0182
- D (Experimental)
  Interventions: Drug: placebo; Drug: NNC 0070-0002-0182

INTERVENTIONS:
Drug: NNC 0070-0002-0182 — 4mg initial dose (12 subjects active; 3 subjects placebo); 2mg weekly maintenance dose; for s.c. injection 20mg/vial
  Arms: A
Drug: placebo — Placebo for s.c. injection
Drug: NNC 0070-0002-0182 — 12mg initial dose (12 subjects active; 3 subjects placebo); 6mg weekly maintenance dose; for s.c. injection 20mg/vial
  Arms: B
Drug: NNC 0070-0002-0182 — 32mg initial dose (12 subjects active; 3 subjects placebo); 16mg weekly maintenance dose; for s.c. injection 20mg/vial
  Arms: C
Drug: NNC 0070-0002-0182 — 60mg initial dose (12 subjects active; 3 subjects placebo); 30mg weekly maintenance dose; for s.c. injection 20mg/vial
  Arms: D

SUMMARY:
This trial will be conducted in the United States of America (USA). The aim of the trial is to investigate whether the drug is safe, well tolerated and to investigate the efficacy of NNC 0070-0002-0182 for the treatment of obesity. The subjects will be treated with drug and placebo. This registration covers the phase 2 part of a combined phase 1/phase 2 trial (phase 1 part of trial conducted between November 2007 and April 2008).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 30.0-39.0 kg/m2 (obese)
* Females who consent to using double barrier method of contraception, are post-menopausal and older than 50 years, or have had total hysterectomy

Exclusion Criteria:

* Clinically significant diseases
* Blood pressure greater than 140/90 mmHg
* Evidence of depression
* Recent diet attempts, treatment with diet drugs (within 3 months)
* Liposuction or other surgery for weight loss within the last year
* Evidence of eating disorders (bulimia, binge eating)
* Restricted diets (Kosher, vegetarian)
* Smoker or history of drug or alcohol abuse
* Females of childbearing potential: positive pregnancy test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2007-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of NNC 0070-0002-0182 multiple doses | after 6 weeks

SECONDARY OUTCOMES:
Pharmacokinetics of NNC 0070-0002-0182 and its isomer | at 8 weeks
Assessment of changes in food consumption and hunger | at 6 weeks
Change in weight, waist and hip measurements and mood | at 6 weeks
Change in body composition and resting metabolism | at 6 weeks
Intervention arm D only: Change in insulin sensitivity (HOMA) | at 6 weeks
Intervention arm D only: Change from baseline in body fat (DEXA) | at 6 weeks
Intervention arm D only: Change from baseline in indirect calorimetry | at 6 weeks
Intervention arm D only: Change from baseline in adiponectin, hsCRP | at 6 weeks
Intervention arm D only: Antibody assessment | at 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- United States (2):
  - Novo Nordisk Investigational Site, Evansville, Indiana
  - Novo Nordisk Investigational Site, Madison, Wisconsin

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com